CLINICAL TRIAL: NCT05397184
Title: Phase 1 Study of Base Edited CAR7 T Cells to Treat T Cell Malignancies (TvT CAR7)
Brief Title: Base Edited CAR7 T Cells to Treat T Cell Malignancies (TvT CAR7)
Acronym: TvT CAR7
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: UCL Great Ormond Street Institute of Child Health (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19IC17
Record Dates: First submitted 2022-05-13; First posted 2022-05-31 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Relapsed/Refractory T-cell Acute Lymphoid Leukaemia
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Intervention Model Description: Phase 1, open label, non randomised
Masking Description: Not applicable (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-dose intravenous infusion of a banded dose of CAR7+ T cells/kg BECAR7 (Experimental): Single-dose intravenous infusion (weight-based dosing) of CAR7+ T cells/kg BECAR7 Total duration of treatment: 28 days Follow-up: 12 months Patients will undergo careful screening to confirm that this treatment is adequate for them. Chemotherapy will be given prior to BE CAR-7 infusion. Patients will then receive a single infusion of the BE CAR-7 cells and will be closely monitored in hospital via blood and bone marrow tests for safety and to check the levels of BE CAR-7 and leukaemia cells. Patients are expected to be in hospital for 4-6 weeks for the BE CAR-7 therapy and the transplant will be scheduled 2-4 weeks after the end of BE CAR7 if leukaemia cells are no longer detectable. Patients will be monitored on the study for 1 year every month for the first 3 months and then every 6 months and then long term in routine clinics.
  Interventions: Biological: Cryopreserved BE CAR7 T cells (BE752TBCCLCAR7PBL)

INTERVENTIONS:
Biological: Cryopreserved BE CAR7 T cells (BE752TBCCLCAR7PBL) — Single-dose intravenous infusion (weight-based dosing) of a banded dose of CAR7+ T cells/kg BECAR7 Total duration of treatment: 28 days Follow-up: 12 months
  Other Names: BECAR7

SUMMARY:
T-cell leukaemia is an uncommon type of blood cell cancer that affects white blood cells (T cells). This phase I clinical trial will treat children aged 6 months up to 16 years with T cell leukaemia which has come back (relapsed) after chemotherapy or is not responding to chemotherapy (refractory). The cell therapy is made from white blood cells (T cells) collected from a healthy donor and changed so they can kill other T cells, including leukaemia cells. These 'ready-made' CAR T cells have been made using a new technique called CRISPR base editing to modify them DNA code and have been given the name BE CAR-7. This technique allows them to work after chemotherapy and also disarms them to prevent effects against normal cells. The main aim of this study is to assess the safety of the BE CAR-7 treatment and to see if ready-made CAR T cells can eradicate T cell leukaemia ahead of a planned bone marrow transplant.

DETAILED DESCRIPTION:
Who can participate? Patients aged 6 months to 16 years with relapsed/refractory T cell leukaemia ahead of a planned bone marrow transplant

What does the study involve? Patients will undergo careful screening to confirm that this treatment is adequate for them. Chemotherapy will be given prior to BE CAR-7 infusion to improve the ability of T-cells to establish and grow. Patients will then receive a single infusion of the BE CAR-7 cells and will be closely monitored in hospital. Patients are expected to be in hospital for 4-6 weeks for the BE CAR-7 treatment and the transplant will be scheduled 2-4 weeks after the end of BE CAR7 if leukaemia cells are no longer detectable. Patients will be monitored on the study for 1 year after transplant and then long term in routine clinics.

What are the possible benefits and risks of participating? Taking part in the study of testing 'ready-made' CAR T cells could help reduce the amount of disease and get the patient into remission before a bone marrow transplant. Leukaemia is less likely to come back after a bone marrow transplant if levels in the bone marrow are undetectable. The ready-made CAR T cells are being used to try and improve the chances of successful transplantation. Side effects may include low blood cell counts, infections, cytokine storm (severe immune reaction), graft versus host disease (where the donated cells attack the body) and other complications.

ELIGIBILITY:
Demographic characteristics:

1. Male or female patients
2. Age ranging between 6 months and <16 years

Medical and therapeutic criteria:

1. Relapsed/refractory T cell malignancy ahead of planned allogeneic haematopoietic stem cell transplantation (allo-SCT). Morphologically confirmed with leukemic blasts in the bone marrow (>5%) or a quantifiable MRD load (by multiparameter flow cytometry and/or quantitative polymerase chain reaction)
2. CD7+ (>99%) leukaemia associated immunophenotype (LAIP)
3. Eligible and fit for allogeneic hematopoietic stem cells transplantation with suitable donor available
4. Estimated life expectancy ≥12 weeks
5. Lansky (age <16 years at the time of assent/consent) or Karnofsky (age ≥16 years at the time of assent/consent) performance status ≥70; Eastern Cooperative Oncology Group ECOG performance status < 2

Exclusion Criteria:

1. Patients/parents unwilling to undergo a follow-up for 15 years
2. Foreseeable poor compliance to the study procedures
3. Evidence of disease progression after cytoreduction
4. Uncontrollable CNS leukaemia or neurological symptoms defined as CNS grade 3 (per National Comprehensive Cancer Network guidelines)
5. Absence of suitable HLA matched or mismatched donor
6. Weight <6 kg
7. Presence of donor-specific anti-HLA antibodies directed against BE-CAR7
8. GvHD requiring systemic therapy
9. Systemic steroid therapy prednisolone >0.5 mg/kg/day
10. Known hypersensitivity to any of the test materials or related compounds
11. Active bacterial, fungal or viral infection not controlled by standard of care anti-microbial or anti-viral treatment. Uncontrolled bacteraemia/ fungaemia is defined as the ongoing detection of bacteria/fungus on blood cultures despite antibiotic or antifungal therapy. Uncontrolled viraemia is defined as rising viral loads on two consecutive occasions despite antiviral therapy.
12. Risk of pregnancy or non-compliance with contraception (if applicable). Girls of childbearing potential must have been tested negative in a pregnancy test within 14 days prior to inclusion.
13. Lactating female participants unwilling to stop breastfeeding
14. Prior CAR therapy known to be associated with ≥Grade 3 cytokine release syndrome (CRS) or ≥Grade 3 drug-related CNS toxicity

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Frequency and description of adverse events after BE-CAR7 infusion | 1 year
  Incidence of Grade 3-5 toxicities occurring from infusion up to one year follow-up.
  Severe Adverse Reactions of special interest will be CRS, ICANS and GvHD. American Society of Bone Marrow Transplantation grading scales for CRS/ICANS and National Institute of Health criteria for GVHD will be applied. Commo Terminology Criteria nomenclature will be used to grade other adverse events.

SECONDARY OUTCOMES:
Number of patients achieving disease remission ahead of allo-SCT | 28 days
  Remission rate will be assessed by bone marrow and CNS evaluation after 28 days. Disease remission is defined as morphological complete remission (CR) or complete remission with incomplete hematologic recovery (CRi) with MRD <10e-3 by flow and/or PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Waseem Qasim, Professor, Principal Investigator — Great Ormond Street Hospital
Locations (1):
- Ilyas Ali, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No